CLINICAL TRIAL: NCT01886144
Title: Effectiveness of Decompressive and Stabilizing Knee Bracing in Individuals With Unicompartment Knee Osteoarthritis
Brief Title: Effects of Bracing on Knee Osteoarthritis (OA)
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Collaborators: Townsend Design (Unknown)
Responsible Party: Sponsor
Other Study IDs: 402877
Record Dates: First submitted 2013-04-18; First posted 2013-06-25 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Knee Osteoarthritis
Keywords: OA; arthritis; knee OA
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee OA: People with knee OA of one knee
  Interventions: Device: Knee OA Brace

INTERVENTIONS:
Device: Knee OA Brace
  Other Names: Rebel Reliever by Townsend Design

SUMMARY:
Knee osteoarthritis (OA) is characterized by complaints of knee pain, aching and stiffness that commonly alter the way one will climb stairs and walk reducing an individual's function and the activities they may perform on a day-to-day basis. Providing a person with a knee brace designed for OA can help unload the arthritic part of the knee, thereby reducing pain and lead to improved function. The purpose of this study is to determine if use of the Rebel Reliever knee brace manufactured by Townsend Design can reduce pain and stiffness, improve strength and balance, and enhance functional activities such as stair and level gait, and ultimately lead to increased participation in the community.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged between 35 and 70
* Present with diagnosed unicompartment osteoarthritis of the knee

Exclusion Criteria:

* Severe cardiac or pulmonary disease that limits ability to walk.
* Presence of hip, ankle or foot OA or other lower limb pathology that limits ability to walk.
* Bilateral knee OA
* Previous use of an OA knee brace
* Surgical procedure in either leg within the past 6-months
* Anthropometrics that are incongruent with manufacturer's specifications for the Rebel Reliever

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are currently living with Knee OA of one leg
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Score (KOOS) | Baseline, 1 week, 2 week, 2 months, 3 months, 6 months
Change in Adductory knee force during stair climbing | Baseline, 2 weeks, 2 months

SECONDARY OUTCOMES:
Change in 6 Minute Walk Test | Baseline, 2 weeks, 2 months
Change in Balance | Baseline, 2 weeks, 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lamberg, EdD, PT, Principal Investigator — Stony Brook Univ
Locations (1):
- Stony Brook University; Rehabilitation Research and Movement Performance (RRAMP) Laboratory, Stony Brook, New York, United States